CLINICAL TRIAL: NCT03484793
Title: Using Big Data and Deep Neural Network to Prevent Medication Errors
Brief Title: Reduce Medication Errors by Translating AESOP Model Into CPOE Systems
Acronym: AESOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Taipei Medical University Shuang Ho Hospital (Other); Taiwan College of Healthcare Executives (Unknown); Taipei Medical University Taipei Municipal Wan Fang Hospital (Unknown); Case Western Reserve University (Other); Cardinal Tien Hospital (Other); Yong He Cardinal Tien Hospital (Unknown); Chang Hua Christian Hospital (Unknown); Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NSC105-2634-F-038-001
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: AESOP Model; Big data; medication error; data mining; patient safety; CPOE; CDSS; alarm fatigue; association rule mining.
MeSH Terms: conditions — Hypertension; Alert Fatigue, Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AESOP integrated to CPOE for reducing medication errors (Experimental): 18 were assigned to the experimental group
  Interventions: Other: AESOP service system
- Non AESOP (No Intervention): 19 were assigned to the traditional CPOE system

INTERVENTIONS:
Other: AESOP service system — Investigators develop an electronic reminder in CPOE system which notifies physicians when there appears to be an inappropriate prescription. At the time, a physician saves a typed prescription, our system analyzes the patient's medications, diseases and uses the knowledge base to determine whether a medication is uncommonly prescribed to all diseases in a given prescription. If the system detects the common associations of medications and diseases in a given prescription, it considers an appropriate prescription, and, if not, an actionable reminder is shown onscreen. To the right of each suggested uncommon medication is a reason why the reminder is appearing. Physicians can accept the reminder or ignore the reminder.
  Arms: AESOP integrated to CPOE for reducing medication errors

SUMMARY:
Medication errors are common, life-threatening, costly but preventable. Information technology and automated systems are highly efficient for preventing medication errors and therefore widely employed in hospital settings. In this study, investigators would perform a cluster randomized controlled trial of a clinical reminding system that uses DNN and Probabilistic models to detect and notify physicians of inappropriate prescriptions, giving them the opportunity to correct these gaps and increase prescriptions completeness. This study aim is to assess whether or not this system would improve prescription notation for a broad array of patient conditions.

DETAILED DESCRIPTION:
This paper focuses on "Big data" in the knowledge base, using "Data minig" study of DM (Disease-Medication) and MM (Medication-Medication) of relevance to develop associated decision resources system-"the intelligent safety system" (Advanced Electronic Safety of Prescriptions,AESOP Model), and test the system in the clinical environment in hospital can assist physicians when open orders reduce medication errors, the system is named "AESOP Model".

ELIGIBILITY:
Inclusion Criteria:

* Physicians who are working at the outpatient clinics in hospitals.
* Physicians who sign the consent form

Exclusion Criteria:

* Physicians who are unable to participate in this trial for the whole process
* Physicians who do not sign the consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The acceptance rate of reminder between two groups intervention and control | 3 months
  The primary outcome of this study is the acceptance rate of the reminder, defined as the number of reminders accepted divided by number of unique reminders presented. In certain instances, physicians might see the same reminder serially, so we aggregate presentations and acceptance of the same reminder for the same patients' prescriptions in our calculation of the acceptance rate.

SECONDARY OUTCOMES:
The changes in the number of reminder for each group | 3 months
  As a secondary outcome, we measure the number of inappropriate prescriptions rate documented in the two groups during the two time periods and calculate the unadjusted relative rate of inappropriateness notation in the intervention group by comparing the number of inappropriateness recorded in the intervention arm during the intervention period to all other groups. The unadjusted relative rate is defined as the ratio (errorsintervention-post/errorscontrol-post)/ (errorsintervention-pre/errorscontrol-pre).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan MD Li, PhD, Study Chair — Taipei Medical University; Chuya Huang, MA, Study Director — Taipei Medical University
Locations (1):
- TMU-Shuang-Ho Hospital, Taipei, Taiwan